CLINICAL TRIAL: NCT05569616
Title: Investigation of the Effect of Hand Massage and Play Activity on Loneliness, Comfort and Psychological Well-Being Levels in the Elderly
Brief Title: Hand Massage and Play Activity in the Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, AYSUN KAZAK, Lecturer, Mersin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AKAZAK.TEZ-KTÜ
Record Dates: First submitted 2022-09-28; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Nursing Caries
Keywords: Hand massage Play activity Psychological well-being Elderly

STUDY DESIGN:
Intervention Model Description: The research was planned as a pre-test-post-test randomized controlled and single-center study in order to examine the effects of hand massage and play activity on loneliness, comfort and psychological well-being in the elderly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hand massage group (Experimental): Based on the hand massage procedure, hand massage with baby oil will be applied for 20 minutes, three times a week (12 times in total) for 4 weeks.
  Interventions: Other: Hand massage
- Play activity group (Experimental): It will be played in groups of two for one hour once a week. The application will take 4 weeks.
  Interventions: Other: Play activity
- Control group (No Intervention): These elderly people in the control group will benefit from the standard care practices offered in the institution, and no intervention will be given to these elderly people by the researcher.

INTERVENTIONS:
Other: Hand massage — Hand massage is a simple comfort intervention that involves touch and conveys care that can easily be incorporated independently into routine nursing care activities. Hand massage is a western technique that includes five basic classical massage manipulations, including eufluorage, petrissage, friction, tapotman and vibration. Kolcaba et al. (2006) hand massage procedure will be applied with baby oil for 20 minutes, three times a week (12 times in total) for 4 weeks.
  Arms: Hand massage group
Other: Play activity — The number of people for the Jenga game was determined as two people in order to strengthen the social relationship among the elderly and to strengthen their psychomotor skills. Each game will be played with two people. For this reason, the elderly will be divided into five separate groups, two people each.These groups will be played the Jenga game for one hour a week on a certain day of the week, accompanied by the researcher, during the activity hours determined by the nursing home. After the game activity (Jenga) application is completed at the end of the fourth week, the post-test scales will be re-administered to the elderly by the researcher.
  Arms: Play activity group

SUMMARY:
There is no study found that examined the effects of hand massage and play activity on the loneliness, comfort and psychological well-being of the elderly in nursing homes. This study was planned as a pretest-posttest randomized controlled dual center study in order to examine the effects of hand massage and play activity on loneliness, comfort and psychological well-being in the elderly. 60 elderly people living in two nursing homes in Mersin city center will form the sample of the study. The sample will consist of three groups as hand massage group, game activity group and control group. The data were using the "Elderly Information Form", "Standardized Mini-Mental Test", "Loneliness Scale fort he Elderly", "General Comfort Scale", "Warwick-Edinburgh Mental Well-Being Scale", "Hand Massage" and "Play Activity (Jenga) will be collected. Hand massage group will be applied hand massage for 20 minutes for four weeks; the game activity group will play Jenga (game activity) for one hour a week. The control group will receive the institution's standart of care. Frequency, number, mean, Student's test and/or Mann-Whitney U test, ANOVA and/or Kruskal-Wallis test, Chi-square test and/or Correlation Analysis will be used in the analysis of the data. As a result of this research, the effects and benefits of hand massage and play activity on the loneliness, comfort and psychological well-being levels of the elderly living in nursing homes will be determined, and it is anticipated that these effects and benefits will be included in evidence-based guidlines.

ELIGIBILITY:
Inclusion Criteria:

1. Be in the age range of 65-84 years
2. Being literate
3. No visual or hearing impairment
4. Ability to communicate verbally
5. Loss of sensation in the hand, arthritis, phlebitis, inflammation, eczema and fracture, etc. absence
6. Absence of any finger or limb loss
7. A score of 25 and above on the Standardized Mini Mental Test
8. Not having been diagnosed with a mental illness such as Parkinson's, Alzheimer's or major depression
9. Staying in a nursing home for at least three weeks
10. Agreeing to participate in the research

Exclusion Criteria:

1. Being 85 years or older
2. Having sensory problems in the hands
3. Having hand and nail deformities
4. Having an open wound or burn on the hands
5. Loss of limbs in fingers
6. Don't have neuropathy

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Elderly Introduction Form | First day
  In this form, which was created by the researchers by scanning the literature; A total of 14 questions aimed at determining the introductory characteristics of the elderly (age, gender, marital status, education level, occupation, number of children, income level, place of residence, smoking and alcohol use, chronic disease diagnosis, duration, medications used, and length of stay in a nursing home) is located.
Standardized Mini Mental Test | will be applied on the first day. If the Standardized Mini Mental Test result is not 25 points or more, the patient will be excluded.
  The standardized version of the original Mini Mental Test developed by Folstein et al. (1975) by Molloy and Standish (1997) is an easy-to-apply test that provides information about the degree of cognitive impairment. This test consists of "orientation, recording, attention, calculation, reminder, language tests and configuration" sections. Test; It is a test that can be administered by physicians, nurses and psychologists in a short time (10 minutes), outpatient conditions or at the bedside. The test was developed for the purpose of short-term cognitive assessment in the elderly, especially in the examination of delirium or dementia.
Loneliness Scale for the Elderly | First week
  It is a measurement tool developed based on the cognitive behavioral approach. The scale, which has 11 items in total, consists of two sub-dimensions, "Emotional Loneliness" and "Social Loneliness":
Loneliness Scale for the Elderly | Forth week
  It is a measurement tool developed based on the cognitive behavioral approach. The scale, which has 11 items in total, consists of two sub-dimensions, "Emotional Loneliness" and "Social Loneliness":
General Comfort Scale | First week
  The levels of the scale, which was formed by taking the taxonomic structure, which includes three levels and four dimensions that constitute the theoretical components of comfort, as a guide; relief (16 items), relief (17 items) and overcoming problems (15 items). Scale dimensions are; physical dimension (12 items), psychospiritual dimension (13 items), environmental dimension (13 items) and sociocultural dimension (10 items).
General Comfort Scale | Forth week
  The levels of the scale, which was formed by taking the taxonomic structure, which includes three levels and four dimensions that constitute the theoretical components of comfort, as a guide; relief (16 items), relief (17 items) and overcoming problems (15 items). Scale dimensions are; physical dimension (12 items), psychospiritual dimension (13 items), environmental dimension (13 items) and sociocultural dimension (10 items).
Warwick-Edinburgh Mental Well-Being Scale | First week
  Scale, Tennant et al. (2007) in order to determine the mental well-being levels of the people of England. The scale is a one-dimensional, 14-item, 5-point Likert scale. Participants respond as "1 = I do not agree at all, 2 = I do not agree, 3 = I agree somewhat, 4 = I agree, 5 = I completely agree).
Warwick-Edinburgh Mental Well-Being Scale | Forth week
  Scale, Tennant et al. (2007) in order to determine the mental well-being levels of the people of England. The scale is a one-dimensional, 14-item, 5-point Likert scale. Participants respond as "1 = I do not agree at all, 2 = I do not agree, 3 = I agree somewhat, 4 = I agree, 5 = I completely agree).

CONTACTS AND LOCATIONS:
Locations (1):
- Nursing home, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No